CLINICAL TRIAL: NCT07221357
Title: ROSETTA CRC-203: A Blinded, Randomized Phase 2/3 Study of Pumitamig in Combination With Chemotherapy Versus Bevacizumab in Combination With Chemotherapy in Participants With Previously Untreated, Unresectable, or Metastatic Colorectal Cancer
Brief Title: A Study to Evaluate the Safety and Efficacy of Pumitamig in Combination With Chemotherapy Versus Bevacizumab in Combination With Chemotherapy in Participants With Previously Untreated, Unresectable, or Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA266-0003; 2025-523224-45 (Other: EU CT Number); U1111-1325-6505 (Other: UTN)
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Untreated, Unresectable, or Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer (mCRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; IFL protocol; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A1 (Experimental)
  Interventions: Drug: Pumitamig; Drug: FOLFOX; Drug: FOLFIRI
- Arm A2 (Experimental)
  Interventions: Drug: Pumitamig; Drug: FOLFOX; Drug: FOLFIRI
- Arm B (Other)
  Interventions: Drug: FOLFOX; Drug: FOLFIRI; Drug: Bevacizumab
- Arm C (Experimental)
  Interventions: Drug: Pumitamig; Drug: FOLFOX; Drug: FOLFIRI; Drug: CAPOX
- Arm D (Other)
  Interventions: Drug: FOLFOX; Drug: FOLFIRI; Drug: Bevacizumab; Drug: CAPOX

INTERVENTIONS:
Drug: Pumitamig — Specified dose on specified days
  Other Names: BMS-986545; BNT327; PM8002
  Arms: Arm A1; Arm A2; Arm C
Drug: FOLFOX — Specified dose on specified days
Drug: FOLFIRI — Specified dose on specified days
Drug: Bevacizumab — Specified dose on specified days
  Arms: Arm B; Arm D
Drug: CAPOX — Specified dose on specified days
  Arms: Arm C; Arm D

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of pumitamig in combination with chemotherapy versus bevacizumab in combination with chemotherapy in participants with previously untreated, unresectable, or metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria

* Participant must previously untreated, histologically confirmed recurrent or metastatic colorectal adenocarcinoma, not amenable to curative surgery.
* Participant must have no known presence of mismatch repair deficient (dMMR) or microsatellite instability-high (MSI-H) colorectal cancer (CRC) per historical results (a validated test should be used).
* Participant must have no known presence of the gene that encodes the protein B-Raf (BRAF) V600E mutation per local testing.
* Participant must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

Exclusion Criteria

* Participant must not have any untreated known central nervous system (CNS) metastases including brain, leptomeningeal and/or spinal cord compression.
* Participant must not have any prior malignancy active within the previous 2 years, except for locally curable cancers that have been apparently cured and considered to be of low risk of recurrence.
* Participant must not have significant cardiovascular disease, such as myocardial infarction, unstable angina, arterial thrombosis or cerebrovascular accident within 6 months prior to randomization, uncontrolled hypertension (≥ 160 systolic, ≥ 100 diastolic mm Hg) despite optimal medical management, or congenital long QT syndrome.
* Participant must not have prior systemic treatment with an anti-PD-1, anti-programmed death (ligand)-1 (PD-L1), anti-PD-L2, CD137 agonists, or anti-cytotoxic T-lymphocyte associated protein 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathways or chemotherapy.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2030-02-02 (Estimated); Study Completion 2034-03-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) (confirmed complete response (CR) or partial response (PR)) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 per investigator assessment | Up to 5 years
  Phase 2
Progression Free Survival (PFS) by RECIST v1.1 per blinded independent central review (BICR) | Up to 5 years
  Phase 3

SECONDARY OUTCOMES:
PFS by RECIST v1.1 per investigator assessment | Up to 5 years
  Phase 2
Duration of Response (DOR) (CR or PR) by RECIST v1.1 per investigator assessment | Up to 5 years
  Phase 2
Time to Response (TTR) (CR or PR) by RECIST v1.1 per investigator assessment | Up to 5 years
  Phase 2
Disease control (Best Overall Response (BOR) of confirmed CR, confirmed PR, or Stable Disease (SD)) by RECIST v1.1 per investigator assessment | Up to 5 years
  Phase 2
Recommended dose of Pumitamig for Phase 3 | Up to 5 years
  Phase 2
Overall Survival (OS) | Up to 5 years
  Phase 3
OR by RECIST v1.1 per BICR | Up to 5 years
  Phase 3
DOR by RECIST v1.1 per BICR | Up to 5 years
  Phase 3

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (229):
- United States (45):
  - Local Institution - 0432, Springdale, Arkansas
  - Local Institution - 0263, Los Angeles, California
  - Local Institution - 0345, Orange, California
  - Local Institution - 0317, San Francisco, California
  - Local Institution - 0330, Santa Monica, California
  - Local Institution - 0293, Stanford, California
  - Florida Cancer Specialists - East, Cape Coral, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Local Institution - 0269, Tampa, Florida
  - Local Institution - 0276, Duluth, Georgia
  - Local Institution - 0369, Marietta, Georgia
  - Local Institution - 0030, Chicago, Illinois
  - Local Institution - 0433, Chicago, Illinois
  - Local Institution - 0335, Iowa City, Iowa
  - Local Institution - 0262, Baltimore, Maryland
  - Maryland Oncology Hematology - Silver Spring, Silver Spring, Maryland
  - Local Institution - 0471, Boston, Massachusetts
  - Local Institution - 0430, Ann Arbor, Michigan
  - Local Institution - 0254, Grand Rapids, Michigan
  - Local Institution - 0572, Maple Grove, Minnesota
  - Local Institution - 0318, Kansas City, Missouri
  - Local Institution - 0336, St Louis, Missouri
  - Local Institution - 0334, Omaha, Nebraska
  - Northwell Health/ RJ Zuckerberg Cancer Center, Lake Success, New York
  - Local Institution - 0270, Mineola, New York
  - Local Institution - 0273, New Hyde Park, New York
  - Local Institution - 0290, Charlotte, North Carolina
  - Local Institution - 0526, Fargo, North Dakota
  - Local Institution - 0339, Columbus, Ohio
  - Local Institution - 0605, Oklahoma City, Oklahoma
  - Local Institution - 0348, Allentown, Pennsylvania
  - Local Institution - 0604, Pittsburgh, Pennsylvania
  - Local Institution - 0312, Sioux Falls, South Dakota
  - Local Institution - 0333, Nashville, Tennessee
  - Sarah Cannon Institute, Nashville, Tennessee
  - Texas Oncology Dallas Fort Worth West (DFWW) - Arlington Cancer Center North, Arlington, Texas
  - Texas Oncology, PA, Austin, Texas
  - Local Institution - 0252, Houston, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Local Institution - 0426, Salt Lake City, Utah
  - Local Institution - 0278, Fairfax, Virginia
  - Local Institution - 0577, Norfolk, Virginia
  - Local Institution - 0491, Edmonds, Washington
  - Local Institution - 0253, Seattle, Washington
  - Local Institution - 0578, Vancouver, Washington
- Argentina (5):
  - Local Institution - 0071, ABB, Buenos Aires F.D.
  - Local Institution - 0174, Buenos Aires
  - Local Institution - 0073, Buenos Aires
  - Local Institution - 0069, Buenos Aires
  - Local Institution - 0172, Buenos Aires
- Australia (14):
  - Local Institution - 0277, Liverpool, New South Wales
  - Local Institution - 0157, St Leonards, New South Wales
  - Local Institution - 0274, Birtinya, Queensland
  - Local Institution - 0215, Herston, Queensland
  - Local Institution - 0191, Woolloongabba, Queensland
  - Local Institution - 0156, Adelaide, South Australia
  - Local Institution - 0155, Elizabeth Vale, South Australia
  - Local Institution - 0196, Ballarat, Victoria
  - Local Institution - 0190, Epping, Victoria
  - Local Institution - 0194, Shepparton, Victoria
  - Local Institution - 0519, St Albans, Victoria
  - Local Institution - 0154, Perth, Western Australia
  - Local Institution - 0160, Malvern
  - Local Institution - 0159, Wentworthville
- Austria (3):
  - Local Institution - 0078, Linz
  - Local Institution - 0178, Salzburg
  - Local Institution - 0082, Vienna
- Belgium (5):
  - Local Institution - 0103, Edegem, Antwerpen
  - Local Institution - 0179, Brussels, MO
  - Local Institution - 0122, Roeselare, West-Vlaanderen
  - Local Institution - 0118, Brussels
  - Local Institution - 0115, Leuven
- Brazil (7):
  - Local Institution - 0267, Curitiba, Paraná
  - Local Institution - 0331, Natal/RN, Rio Grande do Norte
  - Local Institution - 0342, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0373, Santa Cruz do Sul, Rio Grande do Sul
  - Local Institution - 0266, Barretos, São Paulo
  - Local Institution - 0268, São Paulo
  - Local Institution - 0341, São Paulo
- Canada (6):
  - Local Institution - 0550, Calgary, Alberta
  - Local Institution - 0260, Halifax, Nova Scotia
  - Local Institution - 0255, Ottawa, Ontario
  - Local Institution - 0421, Toronto, Ontario
  - Local Institution - 0258, Montreal, Quebec
  - Local Institution - 0423, Montreal, Quebec
- Chile (3):
  - Local Institution - 0171, Recoleta, Santiago Metropolitan
  - Local Institution - 0463, Santiago, Santiago Metropolitan
  - Local Institution - 0175, Santiago, Santiago Metropolitan
- China (23):
  - Local Institution - 0595, Hefei, Anhui
  - Local Institution - 0499, Chongqing, Chongqing Municipality
  - Local Institution - 0354, Fuzhou, Fujian
  - Local Institution - 0388, Fuzhou Fujian, Fujian
  - Local Institution - 0414, Guangzhou, Guangdong
  - Local Institution - 0130, Guangzhou, Guangdong
  - Local Institution - 0390, Tianjin, Hebei
  - Local Institution - 0353, Harbin, Heilongjiang
  - Local Institution - 0384, Nanyang, Henan
  - Local Institution - 0391, Wuhan, Hubei
  - Local Institution - 0411, Changsha, Hunan
  - Local Institution - 0398, Yangzhou, Jiangsu
  - Local Institution - 0381, Nanchang, Jiangxi
  - Local Institution - 0352, Shenyang, Liaoning
  - Local Institution - 0355, Shenyang, Liaoning
  - Local Institution - 0378, Shanghai, Shanghai Municipality
  - Local Institution - 0498, Chengdu, Sichuan
  - Local Institution - 0360, Hangzhou, Zhejiang
  - Local Institution - 0383, Hangzhou, Zhejiang
  - Local Institution - 0409, Beijing
  - Local Institution - 0457, Hangzhou
  - Local Institution - 0356, Shanghai
  - Local Institution - 0412, Wuhan
- Czechia (4):
  - Local Institution - 0248, Prague, Praha 5
  - Local Institution - 0461, Prague, Praha, Hlavní Mesto
  - Local Institution - 0180, Brno
  - Local Institution - 0188, Hradec Králové
- France (11):
  - Local Institution - 0202, Marseille, Bouches-du-Rhône
  - Local Institution - 0590, Besançon, Doubs
  - Local Institution - 0182, Saint-Herblain, Loire-Atlantique
  - Local Institution - 0125, Nantes, Pays de la Loire Region
  - Local Institution - 0121, Marseille, Provence-Alpes-Côte d'Azur Region
  - Local Institution - 0138, Dijon
  - Local Institution - 0183, Paris
  - Local Institution - 0181, Pessac
  - Local Institution - 0127, Rouen
  - Local Institution - 0097, Toulose
  - Local Institution - 0098, Villejuif
- Germany (15):
  - Local Institution - 0591, Erlangen, Bavaria
  - Local Institution - 0033, Dresden, Saxony
  - Local Institution - 0035, Berlin
  - Local Institution - 0061, Bochum
  - Local Institution - 0588, Chemnitz
  - Local Institution - 0057, Düsseldorf
  - Local Institution - 0040, Frankfurt
  - Local Institution - 0058, Göttingen
  - Local Institution - 0039, Hamburg
  - Local Institution - 0594, Hamburg
  - Local Institution - 0041, Leipzig
  - Local Institution - 0060, Mainz
  - Local Institution - 0059, Mannheim
  - Local Institution - 0034, München
  - Local Institution - 0037, Ulm
- Local Institution - 0203, Veszprém, Hungary
- India (7):
  - Local Institution - 0010, Nashik, Dādra and Nagar Haveli and Damān and Diu
  - Local Institution - 0036, Mumbai, Maharashtra
  - Local Institution - 0552, Mumbai, Maharashtra
  - Local Institution - 0006, Delhi
  - Local Institution - 0554, Delhi
  - Local Institution - 0557, Puducherry
  - Local Institution - 0038, Pune
- Italy (8):
  - Local Institution - 0584, San Giovanni Rotondo, Foggia
  - Local Institution - 0231, Milan, Milano
  - Local Institution - 0227, Catania
  - Local Institution - 0111, Milan
  - Local Institution - 0236, Napoli
  - Local Institution - 0221, Padua
  - Local Institution - 0226, Pisa
  - Local Institution - 0233, Reggio Emilia
- Japan (18):
  - Local Institution - 0053, Chiba, Chiba
  - Local Institution - 0045, Matsuyama, Ehime
  - Local Institution - 0051, Sapporo, Hokkaido
  - Local Institution - 0047, Kobe, Hyōgo
  - Local Institution - 0056, Yokohama, Kanagawa
  - Local Institution - 0476, Kurashiki, Okayama-ken
  - Local Institution - 0066, Suita, Osaka
  - Local Institution - 0521, Takatsuki, Osaka
  - Local Institution - 0046, Hidaka, Saitama
  - Local Institution - 0475, Chuo-ku, Tokyo
  - Local Institution - 0044, Koto-ku, Tokyo
  - Local Institution - 0473, Chikusa-ku
  - Local Institution - 0052, Fukuoka
  - Local Institution - 0493, Kashiwa
  - Local Institution - 0597, Kitaadachi-gun
  - Local Institution - 0506, Osaka
  - Local Institution - 0067, Sendai
  - Local Institution - 0054, Sunto-gun
- Netherlands (4):
  - Local Institution - 0112, Amsterdam, North Holland
  - Local Institution - 0170, Groningen
  - Local Institution - 0216, Tilburg
  - Local Institution - 0167, Utrecht
- Poland (7):
  - Local Institution - 0364, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0452, Jelenia Góra, Lower Silesian Voivodeship
  - Local Institution - 0363, Warsaw, Masovian Voivodeship
  - Local Institution - 0525, Warsaw, Masovian Voivodeship
  - Local Institution - 0359, Warsaw, Masovian Voivodeship
  - Local Institution - 0451, Gliwice, Silesian Voivodeship
  - Local Institution - 0362, Opole
- Romania (6):
  - Local Institution - 0282, Cluj-Napoca, Cluj
  - Local Institution - 0100, Bucharest
  - Local Institution - 0142, Cluj-Napoca
  - Local Institution - 0189, Craiova
  - Local Institution - 0370, Iași
  - Local Institution - 0143, Iași
- Singapore (4):
  - Local Institution - 0145, Singapore, Central Singapore
  - Local Institution - 0147, Singapore
  - Local Institution - 0285, Singapore
  - Local Institution - 0511, Singapore
- South Korea (6):
  - Local Institution - 0406, Seongnam, Gyeonggido
  - Local Institution - 0404, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0394, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0395, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0492, Seoul
  - Local Institution - 0405, Seoul
- Spain (8):
  - Local Institution - 0163, Badalona, Barcelona [Barcelona]
  - Local Institution - 0240, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0229, Madrid, Madrid, Comunidad de
  - Local Institution - 0225, Pamplona, Navarre
  - Local Institution - 0228, Madrid
  - Local Institution - 0232, Málaga
  - Local Institution - 0593, Santiago de Compostela
  - Local Institution - 0234, Seville
- Sweden (3):
  - Local Institution - 0074, Stockholm, Stockholm County
  - Local Institution - 0185, Gothenburg, Västra Götaland County
  - Local Institution - 0400, Lund
- Taiwan (6):
  - Local Institution - 0301, Kaohsiung Niao Sung Dist, Kaohsiung
  - Local Institution - 0289, Kaohsiung City
  - Local Institution - 0291, Tainan, Taiana
  - Local Institution - 0297, Taipei
  - Local Institution - 0300, Taipei
  - Local Institution - 0449, Taoyuan District
- Turkey (Türkiye) (5):
  - Local Institution - 0020, Adana
  - Local Institution - 0065, Ankara
  - Local Institution - 0018, Erzurum
  - Local Institution - 0296, Istanbul
  - Local Institution - 0295, Kadiköy/Istanbul
- United Kingdom (5):
  - Local Institution - 0305, Manchester, Lancashire
  - Local Institution - 0307, Glasgow
  - Local Institution - 0368, Kent
  - Local Institution - 0596, London
  - Local Institution - 0316, Sutton

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07221357.html